CLINICAL TRIAL: NCT02709057
Title: Effect of Lifestyle Intervention on Incident Diabetes in Individuals With Impaired Fasting Glucose and Low or High Genetic Risk for the Development of Type 2 Diabetes
Brief Title: Lifestyle Intervention in Individuals With Low or High Genetic Risk for Type 2 Diabetes
Acronym: T2D-GENE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Eastern Finland (Other)
Responsible Party: Principal Investigator, Markku Laakso, Professor, University of Eastern Finland
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: T2D-GENÈ
Record Dates: First submitted 2016-03-06; First posted 2016-03-15 (Estimated); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Life-style intervention 1 (Active Comparator): Life-style intervention in participants with low genetic risk score: The 3-year lifestyle intervention includes 7-9 group sessions (two additional group sessions for participants whose body mass index exceeds 28 kg/m2) on diet (healthy diet according to Nordic and Finnish nutrition recommendations emphasizing appropriate energy intake, meal frequency, consumption of fruits, vegetables and berries, quality of dietary fat and carbohydrates, including sugar and fiber intake) and physical exercise (brisk walking a minimum of 30 minutes per day at least five days a week or other types of exercise, e.g. cycling, cross-country skiing, housework such as leafs raking, resistance training).
  Interventions: Behavioral: Lifestyle intervention
- Life-style intervention 2 (Active Comparator): Life-style intervention in participants with high genetic risk score: The 3-year lifestyle intervention includes 7-9 group sessions (two additional group sessions for participants whose body mass index exceeds 28 kg/m2) on diet (healthy diet according to Nordic and Finnish nutrition recommendations emphasizing appropriate energy intake, meal frequency, consumption of fruits, vegetables and berries, quality of dietary fat and carbohydrates, including sugar and fiber intake) and physical exercise (brisk walking a minimum of 30 minutes per day at least five days a week or other types of exercise, e.g. cycling, cross-country skiing, housework such as leafs raking, resistance training).
  Interventions: Behavioral: Lifestyle intervention
- Control 1 (No Intervention): No intervention in participants with low genetic risk score
- Control 2 (No Intervention): No intervention in participants with high genetic risk score

INTERVENTIONS:
Behavioral: Lifestyle intervention — Life-style intervention includes 7-9 group sessions (two additional group sessions for participants whose body mass index exceeds 28 kg/m2) on diet (healthy diet according to Nordic and Finnish nutrition recommendations emphasizing appropriate energy intake, meal frequency, consumption of fruits, vegetables and berries, quality of dietary fat and carbohydrates, including sugar and fiber intake) and physical exercise (brisk walking a minimum of 30 minutes per day at least five days a week or other types of exercise, e.g. cycling, cross-country skiing, housework such as leafs raking, resistance training).
  Arms: Life-style intervention 1; Life-style intervention 2

SUMMARY:
The aim of the study is to compare the effect of lifestyle intervention (diet and physical activity) by applying modern approaches to lifestyle changes on the prevention of incident T2DM and the worsening of hyperglycemia in people with high number of T2DM risk alleles and in people with low number of T2DM risk alleles compared to corresponding control groups.

DETAILED DESCRIPTION:
AIM: The aim of the study is to compare the effect of lifestyle intervention (diet and physical activity) by applying modern approaches to lifestyle changes on the prevention of incident type 2 diabetes (T2DM) and the worsening of hyperglycemia in people with high number of T2DM risk alleles and in people with low number of T2DM risk alleles compared to corresponding control groups.

STUDY GROUPS. A total of 600 participants will be selected from the METabolic Syndrome In Men (METSIM) study. They are divided into two groups: a) high genetic risk for T2DM on the basis of the genetic risk score (N=300), and b) low genetic risk score for T2DM on the basis of the genetic risk score (N=300). For both of these groups a corresponding control group (N=300) will be selected.

PROTOCOL. 1) The first visit at entry (visit 1) for both intervention and control groups: an interview about physical activity at work and leisure time, smoking, alcohol use, education, occupation, diet, history of medication; clinical measurements: blood pressure, body weight, height, bioimpedance; laboratory measurements including an oral glucose tolerance test, fasting measurements (HbA1c, total cholesterol, HDL cholesterol, total triglycerides, ALT, GAD antibodies); 2) Group sessions (about 15 participants in each) 1-7 described below for the intervention group but not for the control group, 3) A 6 month and 24 month visits (identical to visit 1) for the intervention group but not for the control group; 4) A 3-year visit for both intervention and control groups (identical to visit 1).

Detailed protocol for the intervention group: Dietary guidance in the intervention group is based on the Nordic and Finnish nutrition recommendations and they emphasize appropriate energy intake, meal frequency, consumption of fruits vegetables and berriers, quality of dieatry fat and cardohydrates, including sugar and fiber intake. During the intervention the goals for nutrient and food intake (healthy diet) are: Vegetables, fruits and berries >= 500 g/day, carbohydrates 45-60 E%, sucrose < 10 E%, fiber >=35 g/day, fat 25-40 E%, saturated fat < 10 E%, unsaturated fat >= 2/3 of total fat E%, monosaturated fat 10-20 E%, polysaturated fat 5-10 E%, n-3 fatty acids >= 1E%. The goal for physical activity is brisk walking a minimum of 30 min/day at least five days a week. Walking could be replaced by other types of exercise (e.g. cycling, crioss-country skiing, resistance training, and housework such as leaft raking);

The first year of the intervention will be the most active and includes 4-6 group sessions depending on participants' needs. Group sessions for the intervention group:

Session1 (month 1): Motivation and a 4-day food record and personal feedback from food records to participants.

Sessions 2 and 3 (month 1-2): Healthy dietary pattern and physical activity (see above) Sessions 4 and 5 (month 2-3): Dietary advice for weight loss for the participants with BMI > 28 kg/m2.

6 months visit: 4-day food record and personal feedback from food records to participants.

Session 6: month 12: 4-day food record and personal feedback from food records to participants. Advice for healthy diet and physical activity. Adidtionally a measurement of HbA1c; Session 7 (month 24): 4-day food record and personal feedback from food records to participants. Advice for healthy dietary pattern and physical activity and performance of an oral glucose tolerance test and HbA1c.

Final visit at 36 months: An oral glucose toletance test, HbA1c, and food frequency questionnaire for both intervention and control groups.

Thoughout the study the subjects in the intervention groups will be regularly contacted by the researchers via the website in order to ensure that the subjects stay active regarding the intervention. The web portal also enables the distribution of material and makes virtual discussion possible between the participants and clinical nutritionists. Printed material and discussions by phone will be provided to the participants who do not have access to the internet. In order to help the participants recognize their needs for changes in the diet, available tests (e.g. fiber test, sugar test, fat quality test) provided by the Finnish Heart Association and the Finnish Diabetes Association will be used.

ELIGIBILITY:
Inclusion Criteria:

* Participant of the METSIM Study
* Impaired fasting glucose (IFG) at entry (fasting plasma glucose 5.6-6.9 mmol/l) and with (2-hour glucose 7.8-11.0 mmol/l) or without impaired glucose tolerance (2-hour glucose <7.8 mmol/l) and HbA1c < 6.5%.
* Age 50-75 years
* Male
* Body mass index ≥ 25 kg/m2

Exclusion Criteria:

* Age < 50 years or > 75 years
* Body mass index < 25 kg/m2
* Type 1 or type 2 diabetes or isolated impaired glucose tolerance (2-hour plasma glucose < 5.6 mmol/l and 2-hour plasma glucose 7.8-11.0 mmol/l) or HbA1c ≥ 6.5%
* Chronic diseases preventing to participate in the trial

Ages: 50 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2016-04; Primary Completion 2021-04 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Incident diabetes | 3 years
  Incident diabetes is defined by fasting plasma glucose ≥ 7.0 mmol/l or 2-hour glucose in an oral glucose tolerance test ≥ 11.1 mmol/l or HbA1c ≥ 6.5% or drug treatment started for diabetes during a 3-year follow-up.

SECONDARY OUTCOMES:
The change in glucose area under the curve in an oral glucose tolerance test | 3 years
  The glucose area (mmol/l x min) under the curve in an oral glucose tolerance test is calculated on the basis of glucose measurements (mmol/l) at 0, 30 and 120 min. The change in the glucose area under the curve is the difference between the glucose areas under the curve at randomisation and 3-year visits.
The change in insulin secretion during a 3 year follow-up | 3 years
  Insulin secretion is measured by calculating the glucose area under the curve (mmol/l x min, based on the measurement of glucose in mmol/l at 0 and 30 min) divided by insulin area under the curve (based on the measurement of insulin in pmol/l at 0 and 30 min). The change in insulin secretion is the difference between insulin secretion measured at randomisation and 3-year visits.
The change in insulin sensitivity during a 3 year follow-up | 3 years
  Insulin sensitivity is measured by the Matsuda index (mg/dl, mU/L) based on insulin and glucose measurements at 0, 30 and 120 min. The change in insulin sensitivity is the difference between the Matsuda index at randomisation and at 3-year follow-up visits.

OTHER OUTCOMES:
Incident cardiovascular disease | 3 years
  Incident cardiovascular disease is defined as incident fatal or non-fatal myocardial infarction or cardiovascular death or incident non-fatal or fatal stroke

CONTACTS AND LOCATIONS:
Locations (1):
- University of Eastern Finland, Kuopio, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tolonen UK, Lankinen MA, Laakso M, Schwab US. Association of dietary fibre with type 2 diabetes risk is modified by transcription factor 7 like 2 genotype in men with impaired fasting glucose: The T2D-GENE study. Clin Nutr. 2025 Oct;53:262-269. doi: 10.1016/j.clnu.2025.09.002. Epub 2025 Sep 9. PMID 40961511
- [Derived] Schwab U, Lankinen M, Laakso M. Effect of lifestyle intervention on the risk of incident diabetes in individuals with impaired fasting glucose and low or high genetic risk for the development of type 2 diabetes in men: a T2D-GENE trial. Food Nutr Res. 2021 Sep 23;65. doi: 10.29219/fnr.v65.7721. eCollection 2021. PMID 34650392